CLINICAL TRIAL: NCT00566722
Title: Open Label Study of Adalimumab in Subjects Who Have a Sub-optimal Response to Systemic Therapy or Phototherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Marie Rosenfeld, CRM, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-238
Record Dates: First submitted 2007-12-01; First posted 2007-12-04 (Estimated); Results first posted 2010-05-28 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — Participants received an 80 mg adalimumab loading dose by subcutaneous injection at Baseline (Week 0). From Week 1 to Week 15, participants received 40 mg adalimumab by subcutaneous injection every other week.
  Other Names: ABT-D2E7; Humira

SUMMARY:
The objective of this study was to evaluate the safety and efficacy profile of Humira (adalimumab) in patients who had a sub-optimal response to prior systemic therapy. This open-label study was conducted in a patient population of moderate to severe chronic plaque psoriasis patients, which is an approved patient population for adalimumab.

DETAILED DESCRIPTION:
This 16-week multicenter, open-label study was designed to evaluate the efficacy and safety of a loading dose of 80 mg adalimumab, followed by 40 mg adalimumab every other week in the treatment of psoriasis in patients with a sub-optimal response to etanercept, methotrexate (MTX), or Narrow band Ultraviolet - B (NB-UVB).

Approximately 150 participants were planned for 3 sub-studies: 80 participants with sub-optimal response to etanercept, 40 participants with sub-optimal response to MTX, and 30 participants with sub-optimal response to NB-UVB. Actual enrollment was 82 participants with sub-optimal response to etanercept, 41 participants with sub-optimal response to MTX, and 29 participants with sub-optimal response to NB-UVB.

Screening was performed at least 96 hours and no more than 31 days before the Baseline visit (Week 0). A participant who was eligible for the study based on sub-optimal response to one treatment (MTX, NB-UVB, or etanercept) was required to discontinue that treatment within a specified time before first dose of adalimumab (see descriptions of sub-study groups). In addition, if the participant was also receiving another qualifying treatment, he/she was required to have discontinued the other treatment at least 30 days before the Baseline visit (Week 0).

Adalimumab was administered by subcutaneous (SC) injection. At the Baseline Visit (Week 0), all participants received an initial dose of 80 mg adalimumab SC. Every other week (odd-numbered weeks) from Week 1 to Week 15, participants received 40 mg adalimumab SC.

This was a single group assignment study, that is, all participants received the same treatment; however, data were summarized for 3 groups (sub-studies) that were defined by psoriasis treatments participants received before entering this study: methotrexate, etanercept, or narrow-band, ultraviolet-B.

Efficacy was evaluated using the Physician's Global Assessment (PGA) of disease severity, and patient-reported outcomes: Patient's Global Assessment (PTGA) of disease severity, the Psoriasis-related Pruritus Assessment, the Dermatology Life Quality Index (DLQI), a visual analog scale (VAS) for plaque psoriasis and psoriatic arthritis pain, the Medical Outcomes Study (MOS) Sleep Scale, and the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI: SHP).

Serious and nonserious adverse events were summarized by sub-study of participants (suboptimal response to MTX, suboptimal response to NB-UVB, and suboptimal response to etanercept).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic plaque psoriasis with disease duration of at least 6 months
* Sub-optimal response to treatment with etanercept, methotrexate, or narrow-band UVB phototherapy

Exclusion Criteria:

* Prior treatment with adalimumab
* Multiple concomitant therapy restrictions and/or washouts (topicals, ultraviolet, other systemic psoriasis therapies)
* Prior treatment with natalizumab
* Concurrent active skin diseases/infections
* Poorly controlled medical conditions
* History of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease
* History of certain cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin M Okun, M.D., Ph.D., Study Director — Abbott
Locations (25):
- United States (18):
  - Total Skin and Beauty Dermatology Centers, Birmingham, Alabama
  - Dermatology Research of Arkansas, Little Rock, Arkansas
  - Therapeutics Clinical Research, San Diego, California
  - Florida Academic Dermatology Centers, Miami, Florida
  - Peachtree Dermatology Associates, Atlanta, Georgia
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - ORA Clinical Research and Development, Andover, Massachusetts
  - New York University School of Medicine, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Montifiore Medical Center, The Bronx, New York
  - Paddington Testing Co., Philadelphia, Pennsylvania
  - Clinical Partners, Johnston, Rhode Island
  - Radiant Research, Greer, South Carolina
  - Dermatology Treatment & Research Center, PA Research, Dallas, Texas
  - Baylor Research Institute, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Dermatology Associates, Seattle, Washington
- Canada (7):
  - Kirk Barber Research, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - Eastern Canada Cutaneous Research Associates, Halifax, Nova Scotia
  - Dermatrials Research, Hamilton, Ontario
  - K.Papp Clinical Research Inc, Waterloo, Ontario
  - Siena Medical Research, Montreal, Quebec
  - Centre de Rescherche Dermatologique Du Quebec Metropolitain, Québec, Quebec

REFERENCES:
- [Derived] Strober BE, Poulin Y, Kerdel FA, Langley RG, Gu Y, Gupta SR, Okun MM, Papp KA. Switching to adalimumab for psoriasis patients with a suboptimal response to etanercept, methotrexate, or phototherapy: efficacy and safety results from an open-label study. J Am Acad Dermatol. 2011 Apr;64(4):671-81. doi: 10.1016/j.jaad.2010.03.009. PMID 21414495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were previously treated with etanercept, methotrexate (MTX), or narrow-band ultraviolet-B (NB-UVB) and had a sub-optimal response were recruited for participation in the study.
Pre-assignment Details: Participants who were receiving more than 1 of the treatments (etanercept, MTX, NB-UVB) at the time of screening must have discontinued 1 therapy (e.g., MTX) at least 30 days before first dose of adalimumab and must have discontinued the other therapy (e.g., NB-UVB) during a specified time before first dose of adalimumab. See Detailed Description.
Groups:
- Sub-optimal Response to MTX: MTX treatment must have been administered for at least 4 consecutive months prior to Screening, with no treatment interruptions except for toxicity or intolerability. If there had been a treatment interruption due to toxicity or intolerability, the length of treatment interruption could not have exceeded 14 days. If there was more than one treatment interruption due to toxicity or intolerability (regardless of the length of the treatment interruptions), the participant was not eligible. The last dose of methotrexate must have been at least 4 days but not more than 10 days before the first dose of adalimumab. Suboptimal response was defined as a Physician's Global Assessment of mild (2) or worse.
- Sub-optimal Response to Narrow-band Ultraviolet-B: NB-UVB must have been administered for at least 2 consecutive months prior to Screening, with no treatment interruptions except for toxicity or intolerability. If there had been a treatment interruption due to toxicity or intolerability, the length of treatment interruption could not have exceeded 14 days. If there was more than one treatment interruption due to toxicity or intolerability (regardless of the length of the treatment interruptions), the participant was not eligible. The last treatment with NB UV-B must have been at least 4 days but not more than 10 days before the first dose of adalimumab. Suboptimal response was defined as Physician's Global Assessment of moderate (3) or worse.
- Sub-optimal Response to Etanercept: Etanercept treatment must have been administered for at least 6 consecutive months (or at least 3 consecutive months with deterioration of efficacy observed during the 3 months) prior to Screening, with no treatment interruptions except for toxicity or intolerability, at doses of 50 mg every other week, 50 mg every week, or 25 mg every other week. A treatment interruption due to toxicity or intolerability could not have exceeded 14 days. If there was more than one treatment interruption due to toxicity or intolerability, the participant was not eligible. The last dose of etanercept must have been at least 11 days but not more than 17 days before the first dose of adalimumab. Suboptimal response was defined as a Physician's Global Assessment of mild (2) or worse.
Period: Overall Study
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Started | 41 | 29 | 82
Completed | 39 | 24 | 73
Not Completed | 2 | 5 | 9
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Lack of Efficacy | 1 | 2 | 4
Not completed — Did not meet exclusion criteria | 0 | 0 | 2
Not completed — Serious adverse event | 0 | 1 | 0
Not completed — Noncompliant with drug administration | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept | Total
Number analyzed (Participants) | 41 | 29 | 82 | 152
Age Continuous [Mean (Standard Deviation); unit: years] | 47.4 (13.11) | 45.7 (14.60) | 48.3 (13.70) | 47.6 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 35 | 61
  Male | 28 | 16 | 47 | 91
Region of Enrollment [Number; unit: participants]
  United States | 26 | 10 | 70 | 106
  Canada | 15 | 19 | 12 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Physician's Global Assessment (PGA) of Clear (0) or Minimal (1) at Week 16
Description: The PGA is a 6-point scale used to measure the severity of a patient's disease. Plaque elevation, scaling, and erythema are rated from 0= clear (no plaque elevation; no scaling; erythema=hyperpigmentation, pigmented macules, diffuse faint pink or red coloration) to 5=very severe (plaque elevation=very marked; scaling=very coarse; erythema=very severe [extreme red coloration, dusky to deep red coloration]).
Time Frame: Week 16
Population: All participants who received at least 1 dose of adalimumab were included. Nonresponder imputation (PGA of clear or minimal not achieved) was used for missing data.
Measure: Number; unit: Participants
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Number analyzed (Participants) | 41 | 29 | 82
Participants | 25 | 14 | 40

2. Secondary Outcome: Number of Participants Achieving a PGA of Clear (0) at Week 16
Time Frame: Week 16
Population: All participants who received at least 1 dose of adalimumab were included. Nonresponder imputation (PGA of clear [0] not achieved) was used for missing data.
Measure: Number; unit: Participants
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Number analyzed (Participants) | 41 | 29 | 82
Participants | 15 | 6 | 10

3. Secondary Outcome: Number of Participants Achieving at Least 1 Grade of Improvement in PGA at Week 16 Compared to Screening
Time Frame: From Screening to Week 16
Population: All participants who were enrolled and received a dose of adalimumab were included. Non-responder imputation (1 grade of improvement not achieved) was used for missing data.
Measure: Number; unit: Participants
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Number analyzed (Participants) | 41 | 29 | 82
Participants | 32 | 23 | 59

4. Secondary Outcome: Number of Participants Achieving 0 or 1 on Patient's Global Assessment at Weeks 2, 4, and 8
Description: The Patient's Global Assessment of Psoriasis-Severity is a rating of how well their disease is controlled. 0=complete disease control; 1=good disease control; 2=limited disease control; 3=uncontrolled disease.
Time Frame: Weeks 2, 4, and 8
Population: All participants who received at least 1 dose of adalimumab are included. Nonresponder imputation was used for missing data; that is, participants who did not have an evaluation at the time point were assumed to not have achieved a 0 or 1 on the PGA.
Measure: Number; unit: Participants
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Number analyzed (Participants) | 41 | 29 | 82
Participants
  Week 2 | 5 | 0 | 9
  Week 4 | 13 | 7 | 20
  Week 8 | 22 | 13 | 29

5. Secondary Outcome: Dermatology Life Quality Index (DLQI) Total Score
Description: The DLQI has 10 items and 6 subscales: symptoms and feelings (Q 1 and 2), daily activities (Q 3 and 4), leisure (Q 5 and 6), work and school (Q 7), personal relationships (Q 8 and 9), and treatment (Q 10). Participants rate how much their skin problem affected their life in previous week. Responses are 0 (not at all) to 3=very much. DLQI=total of scores for all items; max=30; min=0.
Time Frame: From Screening to Week 4 and Week 16
Population: All participants who received at least 1 dose of adalimumab were included. Last observation carried forward was used for missing data.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Number analyzed (Participants) | 41 | 29 | 80
Change in scores on a scale
  Week 4 | -4.8 (5.89) | -5.2 (5.45) | -3.3 (4.93)
  Week 16 | -7.0 (7.45) | -6.5 (6.44) | -3.8 (5.66)

6. Secondary Outcome: Number of Participants Achieving DLQI Total Score of 0 at Week 4 and Week 16
Description: DLQI total score of 0 indicates psoriasis had no effect at all on participant's life.
Time Frame: Week 4 and Week 16
Population: All participants who received at least 1 dose of adalimumab were included. Nonresponder imputation (score of 0 not achieved) was used for missing data.
Measure: Number; unit: Participants
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Number analyzed (Participants) | 41 | 29 | 82
Participants
  Week 4 | 6 | 2 | 2
  Week 16 | 12 | 6 | 17

7. Secondary Outcome: Psoriasis-related Pruritus Assessment
Description: The Psoriasis-related Pruritus Assessment is a scale for evaluating pruritus-related to psoriasis over the previous week; values range from 0 (no itching) to 10 (severe itching). A decrease in score indicates an improvement in pruritus.
Time Frame: From Screening to Week 16
Population: All participants who received at least 1 dose of study drug were included. Last observation carried forward was used for missing data.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Number analyzed (Participants) | 41 | 29 | 81
Change in scores on a scale | -2.9 (3.90) | -3.0 (2.96) | -1.7 (3.24)

8. Secondary Outcome: Visual Analog Scale (VAS) for Pain Involving Psoriatic Plaques and/or Psoriatic Arthritis
Description: The participant rates his/her pain during the previous week on a 100 mm VAS, from 0=no pain to 100=pain as bad as it could be. A decrease in score indicates improvement.
Time Frame: From Screening to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Number analyzed (Participants) | 41 | 29 | 81
Change in scores on a scale | -14.7 (24.41) | -21.4 (30.01) | -12.7 (29.90)

9. Secondary Outcome: Percent Work Time Missed Due to Psoriasis
Description: Work and activity impairment due to psoriasis were evaluated using the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI-SHP), a 6-item questionnaire that measures effect of psoriasis on number of hours worked and the number of hours missed from work. It also measures the effect on productivity and regular activities: 0=no effect on work/daily activities; 10=psoriasis prevented me from working/doing daily activities. Decreases in values on each part indicate improvement. At Screening, percent time missed in the previous week ranged from 0% to 40%.
Time Frame: From Screening to Week 16
Population: All participants who received at least 1 dose of adalimumab are included. Last observation carried forward was used for missing data. Screening data were not available for all participants.
Measure: Mean (Standard Deviation); unit: Change in percent time missed
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Number analyzed (Participants) | 25 | 13 | 52
Change in percent time missed | 0.7 (3.43) | 1.3 (4.75) | -0.1 (1.85)

10. Secondary Outcome: Percent Overall Work Impairment Due to Psoriasis
Description: Percent overall work impairment was evaluated using the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI-SHP) (described above). At Screening, overall impairment ranged from 0% to 94%. A decrease in percent overall work impairment indicates improvement.
Time Frame: From Screening to Week 16
Population: All participants who received at least 1 dose of adalimumab were included. Last observation carried forward was used for missing data. Screening data were not available for all participants.
Measure: Mean (Standard Deviation); unit: Change in % overall work impairment
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Number analyzed (Participants) | 25 | 13 | 52
Change in % overall work impairment | -4.0 (28.06) | -6.4 (19.75) | -2.8 (16.92)

11. Secondary Outcome: Percent Impairment While Working Due to Psoriasis
Description: Percent impairment while working was evaluated using the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI-SHP), described above. At Screening, impairment while working ranged from 0% to 90%. A decrease in percent impairment indicates improvement.
Time Frame: From Screening to Week 16
Population: All participants who received at least 1 dose of study drug were included. Last observation carried forward was used for missing data. Screening data were not available for all participants.
Measure: Mean (Standard Deviation); unit: Change in % impairment while working
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Number analyzed (Participants) | 29 | 15 | 59
Change in % impairment while working | -5.5 (30.31) | -8.0 (19.35) | -1.5 (18.46)

12. Secondary Outcome: Percent Activity Impairment Due to Psoriasis
Description: Percent impairment in regular activities was evaluated using the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI-SHP), described above. At Screening, activity impairment due to psoriasis ranged from 0% to 90%.
Time Frame: From Screening to Week 16
Population: All participants who received at least 1 dose of adalimumab were included. Last observation carried forward was using for missing data. Screening data were not available for all participants.
Measure: Mean (Standard Deviation); unit: Change in percent activity impairment
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Number analyzed (Participants) | 40 | 27 | 79
Change in percent activity impairment | -13.3 (33.08) | -12.2 (25.62) | -4.7 (23.03)

13. Secondary Outcome: Sleep Problems Index II
Description: Sleep Problems Index of the Sleep Scale from the Medical Outcomes Study reflects sleep disturbance, perceived sleep adequacy, daytime somnolence, and awakening short of breath or with headache. Participant rates each item from "none of the time" to "all of the time" for the previous 4 weeks. Scores are transformed to 0 to 100 scale; lower scores indicate less impairment. Decrease in score indicates improvement.
Time Frame: From Screening to Week 16
Population: All participants who received at least 1 dose of study drug were included. Last observation carried forward was used for missing data. Screening data were not available for all participants for all items; as a result, not all participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Number analyzed (Participants) | 40 | 27 | 79
Change in scores on a scale | -9.7 (18.01) | -7.7 (15.82) | -2.0 (14.57)

ADVERSE EVENTS:
Time Frame: 26 weeks
Description: Treatment-emergent AEs (TEAEs) were defined as any event with an onset date that was after the first dose of study drug and an onset date no more than 70 days (10 weeks) after the last dose of study drug. The treatment period was 16 weeks and the follow-up period was 10 weeks.
Arm/Group | Sub-optimal Response to MTX | Sub-optimal Response to Narrow-band Ultraviolet-B | Sub-optimal Response to Etanercept
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/29 | 4/82
Other Adverse Events (participants affected / at risk) | 19/41 | 12/29 | 20/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sub-optimal Response to MTX (N=41) | Sub-optimal Response to Narrow-band Ultraviolet-B (N=29) | Sub-optimal Response to Etanercept (N=82)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Diverticulitis Meckel's (Congenital, familial and genetic disorders) | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Helicobacter pylori identification test positive (Investigations) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sub-optimal Response to MTX (N=41) | Sub-optimal Response to Narrow-band Ultraviolet-B (N=29) | Sub-optimal Response to Etanercept (N=82)
Glaucoma (Eye disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 2
Injection site erythema (General disorders) | 3 | 1 | 1
Injection site haemorrhage (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 0
Injection site reaction (General disorders) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0 | 3
Pharyngitis (Infections and infestations) | 0 | 2 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 1 | 5
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 2
Sunburn (Injury, poisoning and procedural complications) | 2 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0
C-reactive protein abnormal (Investigations) | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.